CLINICAL TRIAL: NCT01498367
Title: Renewing Health RCT for the Evaluation of Life-long Tele-monitoring of Patients With Diabetes Mellitus Type 2 in Central Greece
Brief Title: Life-long Tele-monitoring of Patients With Type 2 Diabetes Mellitus in Central Greece
Acronym: RHCluster2GR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Health Authority of Sterea & Thessaly (Other Government)
Collaborators: Ministry for Health and Social Solidarity, Greece (Other); Municipality of Trikala, Greece (Other); e-Trikala S.A. (Industry); Cities Net SA (Industry); Institute of Biomedical Research & Technology, Larissa, Greece (Other); Institute of Communications and Computer Systems, Athens, Greece (Other); Alexander Technological Educational Institute, Thessaloniki, Greece (Other); University of Macedonia, Thessaloniki, Greece (Other); University of Thessaly (Other)
Responsible Party: Principal Investigator, Georgios Koukoulis, Associate Proffesor, Director of the Endocrinology and Metabolic Diseases Department, University Hospital of Larissa, Regional Health Authority of Sterea & Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FR2015; EC Grant Agreement 250487 (Other Grant/Funding Number: European Commission CIP/PSP-ICT Grant Agreement 250487)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Participants in the control group receive usual care. Usual care consists of regular visits to the specialist when required. In the occasion of the visit, HbA1c and glucose measurements are performed and the current oral or insulin therapy is modified if necessary. Patients also receive basic education in the management of diabetes.
- Telemonitoring of diabetes 2 patients (Experimental): Patients will have one educational visit to set up the system and explain how it works. Patients will download their measurements from their tele-glucose meter to their mobile phone and the data will be transferred to the regional database. The care team (a nurse specially trained and the allocated physician) will regularly access the patient's home diary, and will provide the appropriate counselling and medication changes as frequently as necessary. In addition to blood glucose measurements, routine questions about symptoms and eventual difficulties related to diabetes as well as diabetic management will be routinely captured and reported.
  Interventions: Procedure: Telemonitoring of patients with diabetes type 2

INTERVENTIONS:
Procedure: Telemonitoring of patients with diabetes type 2 — Telemonitoring of the patients's blood glucose level measurements using a the tele-glucose meter
  Arms: Telemonitoring of diabetes 2 patients

SUMMARY:
To evaluate whether patients with type 2 diabetes mellitus can be followed by simplified, centralized and large scale tele-monitoring of blood glucose levels and blood pressure, and whether this intervention produces health and economic benefits when introduced without major changes to the existing organization of a large tertiary care center.

DETAILED DESCRIPTION:
The present study aims to examine the clinical and financial effects and the patients' perception and satisfaction of home telemedicine support system for diabetes management versus standard (usual) care. In the intervention group the patients will be provided with a blood glucose meter and a mobile phone and their data will be transferred via the mobile to the regional database and will be assessed by the allocated care team. Appropriate counseling on treatment and symptoms or problems related to diabetes will also be provided.

Measurements of HbA1c will be taken to assess glycaemic control while the dietary and the exercise habits will be assessed by the use of questionnaires. In addition the patients' satisfaction from the use of the telemedicine service will be studied. A Cost-Effective Analysis and Cost Utility Analysis will be applied to evaluate the tele-health service compared with the usual care from the health and social perspective. The effect of the tele-health service in the organization structure of the outpatient hospital department will be evaluated with a qualitative study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 Diabetes
* HbA1c > 53 mmol/mol (7.0 % according to NGSP)
* Capability to use the devices provided
* Being cognitively able to participate
* Capability of filling in questionnaires in german or greek language
* Absence of severe comorbidity prevalent on diabetes with life expectancy < 12 months

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Health related quality of life of the patients measured by the SF-36 version 2 questionnaire | 12 months minimum- at the entry point of the intervention and the end.
HbA1c levels | 12 months minimum - at the entry point and every 3 months.
  Glycated hemoglobin (HbA1c) levels at the entry point and every 3 months (for a period of 12 months minimum)

SECONDARY OUTCOMES:
Emotional functioning in diabetes assessed by the "Problem areas in diabetes questionnaire - PAID © 1999 Joslin Diabetes Center" | 12 months minimum- at the entry point of the intervention and the end.
Physical activity measured by the "International Physical Activity Questionnaire" (IPAQ) | 12 months minimum- at the entry point of the intervention and the end.
Nutrition habits assessed by validated questionnaire. | 12 months minimum- at the entry point of the intervention and the end.
Patients' Acceptance-Satisfaction measured by the WSD Questionnaire | at 2nd and at 12th month
Economic Evaluation (Cost-Effective Analysis- Cost Utility Analysis) | 12 months minimum

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Koukoulis, MD, PhD, Principal Investigator — Endocrinology and Metabolic Diseases Department - Regional University Hospital of Larisa
Locations (1):
- Endocrinology and Metabolic Diseases Department - Regional University Hospital of Larisa, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Polisena J, Tran K, Cimon K, Hutton B, McGill S, Palmer K. Home telehealth for diabetes management: a systematic review and meta-analysis. Diabetes Obes Metab. 2009 Oct;11(10):913-30. doi: 10.1111/j.1463-1326.2009.01057.x. Epub 2009 Jun 16. PMID 19531058
- [Background] Klonoff DC. Diabetes and telemedicine: is the technology sound, effective, cost-effective, and practical? Diabetes Care. 2003 May;26(5):1626-8. doi: 10.2337/diacare.26.5.1626. No abstract available. PMID 12716831
- [Background] Jaana M, Pare G. Home telemonitoring of patients with diabetes: a systematic assessment of observed effects. J Eval Clin Pract. 2007 Apr;13(2):242-53. doi: 10.1111/j.1365-2753.2006.00686.x. PMID 17378871
- See also: "The Renewing Health project is partially funded under the ICT Policy Support Programme (ICT PSP) as part of the Competitiveness and Innovation Framework Programme by the European Community" — http://www.renewinghealth.eu/